CLINICAL TRIAL: NCT03362697
Title: Randomized Clinical Trial on the Safety and Efficacy of Lactobacillus Reuteri DSM 16666/ATCC 55845 & Lactobacillus Reuteri DSM 17938 for Treatment of Pregnant Women With Asymptomatic Bacteriuria or Uncomplicated Acute Cystitis
Brief Title: Lactobacillus Reuteri for Treatment of Uncomplicated UTI in Pregnant Women
Acronym: UTIPregnant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovacion y Desarrollo de Estrategias en Salud (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Pedro Gutierrez Castrellon, Head of Research, Innovacion y Desarrollo de Estrategias en Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUB 0139
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Urinary Tract Infection in Pregnancy
MeSH Terms: interventions — Probiotics; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, double blind allocation concealment, parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization list will by assembled by independient organization not related with participant, care provider, investigators or sponsors. eCRF will include randomization selection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 5*10^8 CFU of Lactobacillus reuteri DSM 16666/ATCC 55845 & Lactobacillus reuteri DSM 17938, PAC-A and Zinc
  Interventions: Dietary Supplement: Probiotics
- Antibiotic (Active Comparator): Amoxicillin + clavulanic acid (500 mg twice daily) for seven days in patients with negative nitrites in dipstick or oral nitrofurantoin (200mg twice per day) for patients with positive nitrates in dipstick
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — The Probiotic group will receive Sachet 1 - contains an instant cranberry drink, consisting of xylitol, monosodium citrate, cranberry aroma, cranberry extract, grape-skin extract, xanthan gum, acesulfame potassium and zinc gluconate and Sachet 2 - contains a total of 5*10^8 CFU of Lactobacillus reuteri DSM 16666/ATCC 55845 & Lactobacillus reuteri DSM 17938, mixed with maltodextrin. Both Sachets should be administered Day 1-14, twice per day This group will also receive for Placebo for Antibiotic treatment day 1-7, twice per day
  Arms: Probiotic
Drug: Antibiotics — Patient in this group will receive for 7 days Amoxicillin + clavulanic acid (500 mg twice daily) for seven days in patients with negative nitrites in dipstick or oral nitrofurantoin (200mg twice per day) for patients with positive nitrates in dipstick. This group will also receive for placebo for probiotics 2 sachets for 14 days
  Arms: Antibiotic

SUMMARY:
Prevalence of uro-genital infections during pregnancy move between 7% to 12% in developed countries, meanwhile in developing countries this figure moved between 14% and until 55%, such is the case of Mexico. Meanwhile use of antibiotics for 3 to 7 days had established as a standard of care, the use of non-antibiotic therapy, such as cranberry powder or probiotics for prevention/treatment of this conditions is scarce. Randomized controlled trial aimed to evaluate the safety and efficacy of probiotic vs. antibiotics to treat pregnant women with uncomplicated cystitis or asymptomatic bacteriuria

DETAILED DESCRIPTION:
Randomized controlled trial, aimed to evaluate the efficacy of Lactobacillus reuteri DSM 16666/ATCC 55845 & Lactobacillus reuteri DSM 17938 for the treatment of pregnant women with asymptomatic bacteriuria or uncomplicated acute cystitis. As primary outcome we will evaluate the number of cases with clinical (symptoms severity) or bacteriological cure in pregnant women with uncomplicated cystitis or asymptomatic bacteriuria after 7 days treatment with probiotics vs. placebo. As secondary outcome we will evaluate a) rate of recurrence cases in each group; b) time to relapse; c) frequency of pyelonephritis; d) birth weight and head circumference; d) number of cases of preterm babies (less than 36 weeks of gestation); e) frequency of antibiotic as rescue treatment; f) frequency of adverse related events in each arm and g) frequency of preeclampsia. Women on active group will receive a combination of at least 5*10^8 CFU of Lactobacillus reuteri DSM 16666/ATCC 55845 & Lactobacillus reuteri DSM 17938, PAC-A and Zinc. Women in control group will receive o Amoxicillin + clavulanic acid (500 mg twice daily) for seven days in patients with negative nitrites in dipstick or oral nitrofurantoin (200mg twice per day) ror patients with positive dipstick.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women on the second or third trimester of pregnancy with positive urine culture according to the operational definition with or without symptoms
* Age 18 to 40 years
* Verbal and Written Informed Consent for participation in the study

Exclusion Criteria:

* Pathologic pregnancy (different for UTI)
* No supplementation of probiotics 2 weeks before study start or during the study period.
* Antibiotic therapy within last 2 weeks before randomization
* Known allergies towards the ingredients of the experimental product
* Inability to comprehend the study protocol
* Systemic diseases
* Multiple pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Clinical and/or Bacteriological cure | 14 days
  Number of cases with improvement of symptoms severity and/or urinary culture during the first seven days of treatment

SECONDARY OUTCOMES:
Recurrence rate | 6 months
  Rate of recurrence cases during the rest of pregnancy
Time to relapse | 6 months
  Time occurred since the finish of treatment until new UTI occurred
Frequency of pyelonephritis | 6 months
  Number of cases of pyelonephritis in each branch
Frequency of preterm babies | 6 months
  Number of children at delivery with <36wekks of gestation
Antibiotic rescue | 6 months
  Use of antibiotics for the treatment of pyelonephritis
Adverse events | 14 days
  Frequency of adverse events in each branch

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nicolle LE. Asymptomatic bacteriuria: when to screen and when to treat. Infect Dis Clin North Am. 2003 Jun;17(2):367-94. doi: 10.1016/s0891-5520(03)00008-4. PMID 12848475
- [Result] Colgan R, Williams M. Diagnosis and treatment of acute uncomplicated cystitis. Am Fam Physician. 2011 Oct 1;84(7):771-6. PMID 22010614
- [Result] Colgan R, Williams M, Johnson JR. Diagnosis and treatment of acute pyelonephritis in women. Am Fam Physician. 2011 Sep 1;84(5):519-26. PMID 21888302
- [Result] Gupta K, Hooton TM, Naber KG, Wullt B, Colgan R, Miller LG, Moran GJ, Nicolle LE, Raz R, Schaeffer AJ, Soper DE; Infectious Diseases Society of America; European Society for Microbiology and Infectious Diseases. International clinical practice guidelines for the treatment of acute uncomplicated cystitis and pyelonephritis in women: A 2010 update by the Infectious Diseases Society of America and the European Society for Microbiology and Infectious Diseases. Clin Infect Dis. 2011 Mar 1;52(5):e103-20. doi: 10.1093/cid/ciq257. PMID 21292654
- [Result] Kazemier BM, Koningstein FN, Schneeberger C, Ott A, Bossuyt PM, de Miranda E, Vogelvang TE, Verhoeven CJ, Langenveld J, Woiski M, Oudijk MA, van der Ven JE, Vlegels MT, Kuiper PN, Feiertag N, Pajkrt E, de Groot CJ, Mol BW, Geerlings SE. Maternal and neonatal consequences of treated and untreated asymptomatic bacteriuria in pregnancy: a prospective cohort study with an embedded randomised controlled trial. Lancet Infect Dis. 2015 Nov;15(11):1324-33. doi: 10.1016/S1473-3099(15)00070-5. Epub 2015 Aug 5. PMID 26255208
- [Result] Romero R, Oyarzun E, Mazor M, Sirtori M, Hobbins JC, Bracken M. Meta-analysis of the relationship between asymptomatic bacteriuria and preterm delivery/low birth weight. Obstet Gynecol. 1989 Apr;73(4):576-82. PMID 2927852
- [Result] Ho M, Chang YY, Chang WC, Lin HC, Wang MH, Lin WC, Chiu TH. Oral Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 to reduce Group B Streptococcus colonization in pregnant women: A randomized controlled trial. Taiwan J Obstet Gynecol. 2016 Aug;55(4):515-8. doi: 10.1016/j.tjog.2016.06.003. PMID 27590374